CLINICAL TRIAL: NCT01714830
Title: The Efficacy of Extracorporal Shock Wave Therapy on Symptoms Relief in Patients With Chronic Non-bacterial Prostatitis / Chronic Pelvic Pain Syndrome
Brief Title: Efficacy of Extracorporal Shock Wave Therapy in Patient With Chronic Non-bacterial Prostatitis / Chronic Pelvic Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farshid Alizadeh, pediatric urologist, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IsfahanUMS1
Record Dates: First submitted 2012-10-12; First posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Extracorporal Shock Wave Therapy; Chronic Non-bacterial Prostatitis; Chronic Pelvic Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham group (Sham Comparator): the same protocol is applied but with the probe being turned off.
  Interventions: Device: turn off standars electromagnetic DUOLITH SD1
- treatment group (Sham Comparator): patients will be treated by ESWT once a week for 4 weeks
  Interventions: Device: standars electromagnetic DUOLITH SD1

INTERVENTIONS:
Device: standars electromagnetic DUOLITH SD1 — In the first group patients will be treated by ESWT once a week for 4 weeks. (Each time 3000 impulses, with 0.25 mJouls/M2 and 3 Hertz of frequency. After each 500 pulses, the probe position will be corrected, using trans-perineal ultrasound.
  Arms: treatment group
Device: turn off standars electromagnetic DUOLITH SD1 — In the control group, the same protocol is applied but with the probe being turned off.
  Arms: sham group

SUMMARY:
Chronic pelvic pain (CPP) can affect both sexes and lasts at least for 3 months. CPP in women could be due to endometrioses, ovarian cyst, colitis, etc, making the correct diagnosis important (1-3). The most prevalent reason for CPP in men is non-bacterial chronic prostatitis and in many cases they are considered equivalent to each other (4).

Chronic non-bacterial prostatitis is associated with pain in pelvic region and could be associated with other symptoms such as dysuria, myalgia, arthralgia, chronic fatigue, burning sensation in the urethra, abdominal, urine frequency, and pain after ejaculation (4-6). Chronic prostatitis / chronic pelvic pain syndrome (CP/CPPS) is devided into two groups: III A Type (inflammatory) and III B (Non-inflammatory). The difference between the two groups is the presence of leukocytes in prostatic secretions after prostate massage, urine and semen (7,8).

In general population, the prevalence of chronic pelvic pain syndrome is about 0.5 percent because many patients do not consider their symptoms as disease, while 6.3% of people may show symptoms (9-11).

One of the most important challenges in the treatment of chronic prostatitis / chronic pelvic pain syndrome, is that its etiology is obscure and it is known as a multi-factorial syndrome. The proposed explanations are infection, psychological reasons, autoimmunity and neuro-myospasm. Hypotheses about endothelial cells defect and cardio vascular disease have also been proposed, upon which the new therapies have been based.

In duplex mapping study of prostatic vessels in two groups of healthy and chronic non-bacterial prostatitis people, it was shown that there was a significant reduction in systolic flow in prostatic arteries in people who had chronic non-bacterial prostatitis, and there was a direct association between pain and blood flow intensity, suggesting chronic ischemia as a possible cause for pain (13). Pain in prostate without significant infection is the hallmark of chronic prostatitis / chronic pelvic pain syndrome (5). In physical exam, prostate or pelvic tenderness may be observed in half of the patients.

The diagnosis of chronic prostatitis / chronic pelvic pain syndrome is challenging. No specific lab test exists for its detection. Prostate specific antigen (PSA) level, which is typically increased in acute infection, is usually normal in this condition. The diagnostic approach in these patients is based on ruling out other curable causes such as benign prostatic hyperplasia or bladder cancer (14-20).

NIH Chronic Prostatitis Symptom Index (NIH-CPSI) is used to evaluate symptom severity and response to treatment in these patients. A reduction of 4-6 points in the score is considered significant response to the treatment (21).

There is no first line treatment for patients of chronic pelvic pain syndrome. The use of anti-bacterial, alpha-blockers or anti-inflammatory drug is logical. However, if the patient does not respond, further administration is not helpful. In non-responders, combination of drugs or other non-medical methods should be considered (23-26).

As discussed earlier, blood flow reduction, ischemia and disorders in endothelium of vessels may cause pain in these patients and methods to improve blow flow may help(13,27). One of these methods is extracorporeal shockwave therapy (ESWT) which is typically used for tendonitis, acceleration in bone reunion and wound healing, improvement in muscle movements through a reduction in passive muscular tonus, increasing muscular range of motion after cerebrovascular accident (CVA), treatment of Peyronie's disease and erectile dysfunction (28-30).

Shoskes et al compared 24 chronic prostatitis patients with 11 controls in terms of vascular stiffness, indexes of increased blood flow, vasodilation and reactive vascular hyperemia, using Endo-PAT ® 2000-Machine. They showed that endothelial disorder and stiffness along with the risk of cardiovascular disorders are increased in CP/CPPS (31).

The use of ESWT for the treatment of CP/CPPS has been evaluated in a few studies. In a double-blind randomized control trial, Zimmermann et al placed 60 patients with chronic pelvic pain syndrome from chronic non-bacterial prostatitis into two groups and treated one of them in 4 sessions with a frequency of 3000 per session. The treatment group showed superior results in terms of symptom improvement(32).

In another study, Zimmermann et al followed 34 patients with chronic pelvic pain syndrome, after one, four and twelve weeks post ESWT in terms of quality of life and pain reduction. They showed that this method is useful and without any complications (33).

Considering the promising results of the cited articles along with the paucity of data in this regard we decided to perform a double-blind sham-controlled study to evaluate the effectiveness of ESWT in CP/CPPS.

DETAILED DESCRIPTION:
Eligible patients will sign an informed consent. Bacterial prostatitis will be ruled out by a 2-glass test (In this method a mid-stream urine sample is collected (10 ml of urine is discarded and the second 10 ml of urine is collected) and then prostate massage is done for a minute by Digital Rectal Exam and then another 10 ml of urine is collected.

After briefing the patients about the method and obtaining written consent from, he will be randomly allocated into either the treatment or control group.

In the first group patients will be treated by ESWT once a week for 4 weeks. (Each time 3000 impulses, with 0.25 mJouls/M2 and 3 Hertz of frequency. After each 500 pulses, the probe position will be corrected, using trans-perineal ultrasound. The used device in this study is the standars electromagnetic DUOLITH SD1- shock waves against erectile dysfunction.

In the control group, the same protocol is applied but with the probe being turned off.

The examination is performed in supine position for patient. For each patient, pelvic pain intensity considering is performed at the beginning and end of study, by VAS. Patients are considered by doctor for NIH index at the beginning and end of study.

Finally, obtained data about pain relief and change in NIH-CPSI are recorded in special profile for each patient and finally are analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Non-addiction to drugs and narcotics.
2. Chronic pelvic pain existence for more than three month and certain diagnosis of chronic non-bacterial / chronic pelvic pain syndrome.
3. Signing an informed consent for treatment by ESWT

Exclusion Criteria:

1. To be under treatment by another method at the beginning of the study
2. Another diagnosis such as prostate cancer is suggested during work-up.
3. Therapy plan alteration.
4. Non-inclination to continue this project.

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
effect of extracorporeal shock wave therapy on pain reduction according to visual analogue scale and NIH-CPSI scale in patients with chronic non-bacterial prostatitis / chronic pelvic pain syndrome | 12 months
  For each patient, pelvic pain intensity considering is performed at the beginning and end of study, by visual analogue scale(VAS). Patients are considered by doctor for NIH index according to NIH-CPSI scale at the beginning and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Alizadeh, pediatric urologist, Principal Investigator — Isfahan University of Medical Sciense